CLINICAL TRIAL: NCT05862038
Title: Biomarkers in Pulsed Field Ablation Versus Cryoballoon Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ana Jordan (Other)
Responsible Party: Sponsor-Investigator, Ana Jordan, Principal investigator, University Hospital Dubrava
Organization: University Hospital Dubrava (Other)
Other Study IDs: KBD01
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study will include consecutive patients undergoing pulsed field ablation (PFA) or cryoballoon (CBA) ablation. Tissue injury and inflammation markers will be measured before and after the procedure.

DETAILED DESCRIPTION:
Study population:

The participants with symptomatic atrial fibrillation scheduled for PFA or CBA procedures Biomarkers of interest: high-sensitive troponin, CRP, NT-proBNP Data collection: Blood samples will be collected at baseline, immediately after the procedure, 24 hours after, and three months after.

Statistical analysis:

Comparisons of biomarker levels between PFA and CBA groups.

Results:

Comparison of biomarker levels between PFA and CBA groups at each time point. Changes in biomarker levels over time within each group. Correlation analysis between biomarker levels and clinical outcomes, such as AF recurrence, LA stiffness, complications, and hospitalization.

ELIGIBILITY:
Inclusion criteria:

* Symptomatic paroxysmal or persistent atrial fibrillation.
* Age between 18 and 75 years.

Exclusion criteria:

* Prior atrial fibrillation ablation.
* History of significant bleeding or thromboembolic events within the last 6 months.
* History of severe renal or liver disease.
* History of malignancy within the last 5 years.
* History of autoimmune disease or immunodeficiency.
* Significant mitral stenosis or other significant valvular heart disease.
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients who are diagnosed with symptomatic paroxysmal or persistent atrial fibrillation and who are scheduled to undergo catheter ablation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
To see if PFA vs CBA increase left atrium stifness by measuring NT-proBNP values after procedures | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ana Jordan, Principal Investigator — University Hospital Dubrava
Locations (1):
- UH Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No